CLINICAL TRIAL: NCT03178643
Title: Enhancing Preventive Therapy of Malaria In Children With Sickle Cell Anemia in East Africa (EPiTOMISE)
Acronym: EPiTOMISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00077428; R01HL134211 (NIH)
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Proguanil; Sulfadoxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Proguanil Oral Tablet (Active Comparator): Proguanil is the current standard of care for chemoprevention of malaria in children with SCA in Kenya. This medication will be taken on a daily basis
  Interventions: Drug: Proguanil Oral Tablet
- Sulfadoxine/Pyrimethanine-Amodiaquine (Active Comparator): Sulfadoxine/Pyrimethanine-Amodiaquine (SP-AQ) is a combination therapy comprised of sulfadoxine and pyrimethamine (two antifolate antimicrobials) co-administered with amodiaquine. This medication is taken on a monthly basis.
  Interventions: Drug: Sulfadoxine/Pyrimethanine-Amodiaquine (SP-AQ)
- Dihydroartemisinin-Piperaquine (DP) (Active Comparator): DP is an artemisinin-combination therapy consisting of the artemisinin derivative dihydroartemisinin and the bisquinoline piperaquine. This medication is taken on a monthly basis.
  Interventions: Drug: Dihydroartemisinin-Piperaquine (DP)

INTERVENTIONS:
Drug: Proguanil Oral Tablet — Dosing of daily proguanil will be approximately 3mg/kg/day,
  Arms: Proguanil Oral Tablet
Drug: Sulfadoxine/Pyrimethanine-Amodiaquine (SP-AQ) — Age 1-5 on Day 1: One tablet 500/25mg SP and one tablet 153mg AQ Day 2 and Day 3: one tablet 153 mg AQ only each day For ages 6-10: Day 1 - 1.5 tablets 500/25mg SP and 1.5 tablets 153mg AQ Days 2 and 3: 1.5 tablets 153mg AQ only each day
  Arms: Sulfadoxine/Pyrimethanine-Amodiaquine
Drug: Dihydroartemisinin-Piperaquine (DP) — 3) The weight-based dosing of tablets of 40/320mg of DP is described below:
  Weight (kg) No. of 40/320mg tabs DP daily for 3 days
  ≤ 5 ¼ 6-10 ½ 11-14 ¾ 15-19 1 20-23 1 ¼ 24-25 1 ½
  Arms: Dihydroartemisinin-Piperaquine (DP)

SUMMARY:
This is a randomized, three-arm, open-label, clinical trial of malaria chemoprevention in children with sickle-cell anemia (SCA) at a single site in Homa Bay, Kenya. The study will enroll 246 children under 10 years of age, randomize participants 1:1:1 to one of three malaria chemoprevention regimens, and follow participants monthly for 12 months in order to record clinical episodes of malaria or SCA-related morbidity. Analyses will compare the efficacy of each regimen to prevent malaria and SCA morbidity.

DETAILED DESCRIPTION:
Purpose of the study:

Primary Objective: To compare the efficacy of daily proguanil with monthly sulfadoxine/pyrimethanine-amodiaquine (SP-AQ) and with monthly dihydroartemisinin-piperaquine (DP) on the incidence of falciparum malaria in children with SCA.

Secondary Objective: To compare the efficacy of these malaria chemoprevention strategies on the incidence of major complications of SCA.

Background & significance

Over 240,000 children with sickle cell anemia (SCA) are born in Africa annually. This number will increase to over 350,000 annual births of children with SCA by the year 2050. Without sophisticated medical care, SCA patients in African settings die at young ages: in a Western Kenya cohort of newborns, 25% of SCA children died before their 3rd birthday. Caring effectively for these children will be a major challenge for developing medical and public health systems in Africa including Kenya, and modeling studies suggest that the adequate provision of effective preventive care can substantially reduce the mortality of these children. Preventive care for SCA children must be evidence-based and tailored to the unique epidemiology of comorbidities in African settings.

Children under 5 years of age in sub-Saharan Africa also suffer the majority of the annual 350 million infections and 500,000 deaths globally. Reducing this burden is a global public health priority, particularly in areas of high transmission like Western Kenya. In the absence of an effective vaccine, global malaria control requires effective treatments and a suite of preventive measures that act upon the parasite, environment, and host. Among these preventive strategies is the administration of prophylactic antimalarials to high risk groups, including pregnant women, infants, and children exposed to seasonal malaria transmission. In these high-risk groups malaria morbidity is substantially reduced by routine periodic intake of effective antimalarials.

Children with SCA are at high risk of life-threatening malaria. In East Africa children with SCA admitted to the hospital with malaria parasites were more likely to die than those without parasites. Malaria is also a precipitant of sickle-cell pain crises, by unclear mechanisms. It remains unclear how SCA influences the overall risk of malaria, because most studies have been hospital based and therefore unsuited to capture mild episodes. The twin observations that malaria is more severe in SCA children and precipitates painful crises in these children indicate that the prevention of P. falciparum infections is critical to prolong the survival of SCA children in malaria-endemic areas.

Design & procedures - This is a randomized, three-arm, open-label, clinical trial of malaria chemoprevention in children with sickle-cell anemia (SCA) at a single site in Homa Bay, Kenya. The study will enroll 246 children under 10 years of age, randomize participants 1:1:1 to one of three malaria chemoprevention regimens, and follow participants monthly for 12 months in order to record clinical episodes of malaria or SCA-related morbidity. Analyses will compare the efficacy of each regimen to prevent malaria and SCA morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 12 months and less than 10 years at enrollment;
* Current attendance at or willingness to attend the study SCA clinic at HBCH;
* Residence in either Homa Bay County or the Rongo or Awendo sub-counties of Migori County;
* Confirmed hemoglobin genotype of HbSS by electrophoresis, HPLC, or PCR;
* No immediate, apparent, or reported plans to relocate residence from Homa Bay County or the Rongo or Awendo sub-counties of Migori County in the next 2 years;
* Ability to take oral medication and be willing to adhere to the medication regimen or caregiver willingness to give the medical regimen as prescribed;
* Ability and willingness of parent or legally authorized representative (LAR) to give informed consent;
* Assent of child in those > 7 years.

Exclusion Criteria:

* Taking routine antimalarial prophylaxis for another indication (including co-trimoxazole for HIV infection);
* Temperature of ≥ 37.5C at screening or history of objective or subjective fever in the preceding 24 hours during screening;
* Known allergy or sensitivity to sulfadoxine, pyrimethamine, amodiaquine, proguanil, dihydroartemisinin, piperaquine, artemether, lumefantrine, pencillin (if under 5 years old), or derivatives of these compounds;
* Known chronic medical condition other than SCA (i.e. malignancy, HIV) requiring frequent medical attention;
* Currently participating in another clinical research study, or having participated in one in the prior 30 days;
* Living in the same household as a previously-enrolled study participant;
* Chronic use of medications known to prolong the QT interval in children (see Appendix J);
* Fridericia's corrected QT interval (QTcF) interval > 450msec.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 246 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Homa Bay County Referral Hospital, Homa Bay Town, Homa Bay County, Kenya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Taylor SM, Korwa S, Wu A, Green CL, Freedman B, Clapp S, Kirui JK, O'Meara WP, Njuguna FM. Monthly sulfadoxine/pyrimethamine-amodiaquine or dihydroartemisinin-piperaquine as malaria chemoprevention in young Kenyan children with sickle cell anemia: A randomized controlled trial. PLoS Med. 2022 Oct 10;19(10):e1004104. doi: 10.1371/journal.pmed.1004104. eCollection 2022 Oct. PMID 36215323

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants will be screened for inclusion in the existing pediatric. Currently, SCA patients are cared for in two parallel clinics: 1) the pediatric medical officer staffs a weekly SCA clinic, and 2) the AMPATH HematoOncology outreach team staffs a monthly 2-day SCA clinic at HBCH.
  Potential participants will be screened for eligibility. If they meet all inclusion criteria and do not meet any exclusion criteria, they will be offered enrollment following informed consent.
Groups:
- Dihydroartemisinin-Piperaquine (DP): DP is an artemisinin-combination therapy consisting of the artemisinin derivative dihydroartemisinin and the bisquinoline piperaquine. This medication is taken on a monthly basis.
  Dihydroartemisinin-Piperaquine (DP): 3) The weight-based dosing of tablets of 40/320mg of DP is described below:
  Weight (kg) No. of 40/320mg tabs DP daily for 3 days
  ≤ 5 ¼ 6-10 ½ 11-14 ¾ 15-19 1 20-23 1 ¼ 24-25 1 ½
Period: Overall Study
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Started | 81 | 83 | 82
Completed | 75 | 67 | 71
Not Completed | 6 | 16 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP) | Total
Number analyzed (Participants) | 81 | 83 | 82 | 246
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 81 | 83 | 82 | 246
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.8 (2.6) | 4.3 (2.3) | 4.7 (2.6) | 4.6 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 36 | 35 | 115
  Male | 37 | 47 | 47 | 131
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Tribe/Ethnic Group: Luo | 80 | 82 | 82 | 244
  Tribe/Ethnic Group: Luhya | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Kenya | 81 | 83 | 82 | 246

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Clinical Malaria Per Patient Year
Description: The primary endpoint is the cumulative incidence of clinical malaria expressed as episodes per person-year at risk. Time at risk will begin when study participants are randomized and receive study drug (i.e. begin chemoprevention) and end when participants reach the end of the observation period.
Time Frame: 12 months
Measure: Number; unit: episodes/patient year
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 81 | 83 | 82
episodes/patient year | 0.04 | 3.05 | 1.36

2. Secondary Outcome: Number of Participants With Severe Anemia
Description: E.g., hemoglobin <5.5 g/dL
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 81 | 83 | 82
Participants | 8 | 9 | 4

3. Secondary Outcome: Number of Participants With Severe Malaria
Description: Positive rapid diagnostic test (RDT).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 81 | 83 | 82
Participants | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Hospitalization for Malaria
Description: Patient admitted to hospital for malaria with confirmed positive RDT.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 81 | 83 | 82
Participants | 3 | 3 | 3

5. Secondary Outcome: Number of Participants With Light Microscopy (LM)-Positive Malaria
Description: LM-positive malaria defined as the reported presence of P. falciparum parasites detected by LM irrespective of RDT or other detection results.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 81 | 83 | 82
Participants | 17 | 11 | 19

6. Secondary Outcome: Number of Participants With Unconfirmed Malaria
Description: Defined as the receipt of antimalarials for suspected malaria episodes that were not confirmed by any objective diagnostic test.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 81 | 83 | 82
Participants | 42 | 25 | 40

7. Secondary Outcome: Number of Participants With Fatal Malaria
Description: Defined as death during hospitalization for malaria with positive RDT.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 81 | 83 | 82
Participants | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Asymptomatic Parasitization
Description: Defined as the presence of parasites during routine follow-up visits as detected by PCR in patients without fever or a history of recent fever.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 81 | 83 | 82
Participants | 45 | 20 | 9

9. Secondary Outcome: Number of Participants With Painful Events
Description: Pain lasting two hours or more without obvious cause.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 81 | 83 | 82
Participants | 33 | 28 | 30

10. Secondary Outcome: Number of Participants With Dactylitis
Description: Pain or tenderness with or without swelling of the hands or feet.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 81 | 83 | 82
Participants | 81 | 57 | 37

11. Secondary Outcome: Number of Participants With Transfusions
Description: Receipt of RBCs (red blood cells) from any caregiver for any indication.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 81 | 83 | 82
Participants | 13 | 7 | 4

12. Secondary Outcome: Number of Participants With Acute Chest Syndrome
Description: Defined as a new pulmonary infiltrate and at least 3 of the following findings: chest pain, temperature elevation > 38.5°C, tachypnea, wheezing, or cough.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 81 | 83 | 82
Participants | 1 | 3 | 0

13. Secondary Outcome: Number of Participants With All-cause Hospitalization
Description: Hospitalization at HBCH or any other inpatient facility with any admitting diagnosis.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 81 | 83 | 82
Participants | 47 | 52 | 40

14. Secondary Outcome: All-cause Deaths
Description: Death by any cause.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 81 | 83 | 82
Participants | 2 | 7 | 1

15. Secondary Outcome: Molecular Markers of Malaria Parasite Drug Resistance
Description: presence of SNPs in parasite genes that confer resistance to the study drugs
Time Frame: 12 months
Population: Data not collected.
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: This protocol collected only SUSARs (Suspected Unexpected Serious Adverse Reactions) and deaths.
Arm/Group | Proguanil Oral Tablet | Sulfadoxine/Pyrimethanine-Amodiaquine | Dihydroartemisinin-Piperaquine (DP)
All-Cause Mortality (participants affected / at risk) | 2/81 | 7/83 | 1/82
Serious Adverse Events (participants affected / at risk) | 22/81 | 22/83 | 19/82
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proguanil Oral Tablet (N=81) | Sulfadoxine/Pyrimethanine-Amodiaquine (N=83) | Dihydroartemisinin-Piperaquine (DP) (N=82)
Painful Crisis (Blood and lymphatic system disorders) | 22 (33) | 22 (28) | 19 (30)
Anemia (Blood and lymphatic system disorders) | 10 (12) | 12 (14) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT03178643/Prot_SAP_000.pdf